CLINICAL TRIAL: NCT04347655
Title: A Novel Approach to the Assessment of the Systemic Circulation and Left Ventricular Performance in Adults
Brief Title: Assessing Systemic Circulation and LV Performance in Adults
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Calgary (Other)
Responsible Party: Principal Investigator, Dr. Satish Raj, Professor of Cardiac Sciences, University of Calgary
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: REB20-0465
Record Dates: First submitted 2020-04-12; First posted 2020-04-15 (Actual); Last update posted 2024-05-08 (Actual); Status verified 2024-05

CONDITIONS: Heart Failure
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Intervention Model Description: Heart Failure Patients (with reduced and preserved ejection fraction) and Healthy Control Subjects will be studied with the same protocol
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- HFrEF (Experimental): patients with heart failure with reduced ejection fraction
  Interventions: Procedure: handgrip test
- HFpEF (Experimental): heart failure with preserved ejection fraction
  Interventions: Procedure: handgrip test
- Control (Active Comparator): healthy (no heart failure) control participants
  Interventions: Procedure: handgrip test

INTERVENTIONS:
Procedure: handgrip test — The patient will be supine for at least 5 minutes to collect baseline data before being handed a dynamometer device. The subject will then be asked to squeeze the dynamometer with maximum force for a minimum of 2 minutes while only engaging their forearm and remaining relaxed in the rest of their body. The subject will then release the dynamometer and remain supine, in recovery, for a minimum of 5 minutes.

SUMMARY:
Background There are significant limitations in the current approaches to assessing 2 important areas of cardiovascular physiology - the systemic circulation and left ventricular (LV) performance. The investigators' have repurposed the concepts of "systemic vascular conductance" to assess systemic circulation, and the "head capacity principle" to assess LV performance. The investigators' now seek to test these concepts in human adults, with heart failure and without heart failure, using non-invasive methods.

Hypothesis There will be a depressed head-capacity curve and reduced power among patients with heart failure which will indicate compromised left ventricular pump function.

Methods The research study will involve a single outpatient visit per subject. The study will take place with the subject supine on a bed/table. The subjects will be instrumented with EKG electrodes and finger blood pressure cuffs. The continuous finger BP device performs a waveform analysis in real-time to determine the non-invasive stroke volume, cardiac output, and blood pressure.

The patient will be supine for at least 5 minutes to collect baseline data before being handed a dynamometer device. The subject will then be asked to squeeze the dynamometer with maximum force for a minimum of 2 minutes while only engaging their forearm and remaining relaxed in the rest of their body. The subject will then release the dynamometer and remain supine, in recovery, for a minimum of 5 minutes.

Following the handgrip test, the instrumentation will be removed and the patient's participation in the study will be complete. The study duration should be about 20 min.

DETAILED DESCRIPTION:
Background There are significant limitations in our current approaches to assessing 2 important areas of cardiovascular physiology - the systemic circulation and left ventricular (LV) performance. Using engineering principles, the investigators' have repurposed 2 concepts to develop novel (and hopefully improved) interpretation of integrated cardiovascular function. These concepts are "systemic vascular conductance" for systemic circulation and the "head capacity principle" for LV performance, which have been demonstrated in animal physiology experiments using a porcine model. In this protocol, the investigators' seek to test these concepts in human adults, with heart failure and without heart failure, using non-invasive methods.

Aims and Hypotheses Primary Aim: To evaluate cardiovascular function in patients with heart failure using a head-capacity relation to assess left ventricular pump function as well as by assessing systemic vascular conductance.

Hypothesis: There will be a depressed head-capacity curve and reduced power among patients with heart failure which will indicate compromised left ventricular pump function. In addition, heart failure patients will have decreased systemic vascular conductance.

Specific Aim#1: The investigators' will compare patients with heart failure with reduced ejection fraction (HFrEF) to healthy (no heart failure) control participants.

Specific Aim #2: The investigators' will compare patients with heart failure with preserved ejection fraction (HFpEF) to healthy (no heart failure) control participants.

Methods The research study will take place in the TRW Building on the University of Calgary Foothills Campus. This will involve a single outpatient visit per subject. Patients can be brought to the TRW building from the Cardiac Function Clinic or Cardiac Device Clinic in a wheelchair, accompanied by a member of the research team or can arrive to the TRW building by their own means. As a part of the consent process, the subject will be asked to allow access to their clinical records for research purposes. This will include collecting information about their heart failure such as their ejection fraction, NYHA class, medications, and whether they have an implanted permanent pacemaker or implanted defibrillator capable of atrial and ventricular pacing.

The study will take place with the subject supine on a bed/table. The subjects will be instrumented with EKG electrodes and finger blood pressure cuffs. The continuous finger BP device performs a waveform analysis in real-time to determine the non-invasive stroke volume, cardiac output, and blood pressure. These will be connected to a laptop for continuous digital acquisition through an analog:digital conversion card.

The patient will be supine for at least 5 minutes to collect baseline data before being handed a dynamometer device. The subject will then be asked to squeeze the dynamometer with maximum force for a minimum of 2 minutes while only engaging their forearm and remaining relaxed in the rest of their body. The subject will then release the dynamometer and remain supine, in recovery, for a minimum of 5 minutes.

Following the handgrip test, the instrumentation will be removed and the patient's participation in the study will be complete. The study duration should be about 20 min.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 years or older
* Clinical heart failure (HFrEF or HFpEF) for heart failure patients and no clinical heart failure for the non-heart failure participants.

Exclusion Criteria:

* Unable or unwilling to provide informed consent
* On intravenous inotrope or pressor medications to maintain their cardiac function

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2021-09-15 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Head-Capacity Curve (HCC) | 1 day
  systolic arterial blood pressure (SBP) when CI = 4 L/min/m2

SECONDARY OUTCOMES:
Cardiac Power | 1 day
  cardiac power (SBP * CI) when CI = 4 L/min/m2
Systemic Vascular Conductance (SVC) | 1 day
  SVC is the slope of the regression line (going through the origin) between SBP and CI

CONTACTS AND LOCATIONS:
Overall Officials: Satish R Raj, MD MSCI, Principal Investigator — University of Calgary
Locations (1):
- University of Calgary, Calgary, Alberta, Canada

IPD SHARING:
Plan to Share IPD: No